CLINICAL TRIAL: NCT02407288
Title: Transcranial Direct Current Stimulation as an add-on Treatment in SSRI-resistant Obsessive Compulsive Disorder : a Randomized Clinical Trial
Brief Title: tDCS as an add-on Treatment in SSRI-resistant OCD
Acronym: TDCSTOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Principal Investigator, BATION Rémy, Dr Rémy Bation, Hôpital le Vinatier
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSR G01
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active tDCS (Active Comparator): patients will received 2 sessions per day for 5 consecutive days. Each session will last 20 minutes. The tDCS device will deliver a direct current of 2mA during 20 minutes. Cathode will be localized in front of the left orbito-frontal on the FP3 point according to the EEG international reference. Anode will be localized in front of the right cerebellum 3 cm below the inion and 1 cm right from the midline
  Interventions: Device: transcranial dirrect current stimulation
- SHAM tDCS (Placebo Comparator): The same procedure will be applied except that the tDCS device will only deliver a current stimulation for the 10 first seconds.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: transcranial dirrect current stimulation — The tDCS device will deliver a direct current of 2mA during 20 minutes. Cathode will be localized in front of the left orbito-frontal on the FP3 point according to the EEG international reference. Anode will be localized in front of the right cerebellum 3 cm below the inion and 1 cm right from the midline
  Other Names: tdcs
  Arms: active tDCS
Device: Sham tDCS
  Arms: SHAM tDCS

SUMMARY:
The purpose of this study is to determine whether tDCS is effective as an add-on treatment in SSRI-resistant patients with obsessive and compulsive disorder

DETAILED DESCRIPTION:
Total number of scheduled patients to be recruited: 46 We used the effect size of the study of Ruffini and colleagues (2009) in which rTMS was used to target the left orbito frontal cortex to calculate the number of patients to be recruited. With a risk alpha of 5%, a power of 80%, the number of patients to be included was 46 with an anticipated rate of 10% of lost to follow-up patients. (calculation was made on the http://www.spc.univ-lyon1.fr/mfcalc/NSN/assistant.htm)

Statistical analysis to address the primary and secondary objectives:

Chi squared test will be applied for quantitative data.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with OCD according to DSM V criteria
* YBOCS score of 16 and above, stable (<20% of variation) during at least one month.
* have received for at least 12 weeks of which 6 weeks was either at the maximum tolerated dose or alternatively the manufacturer's recommended maxi- mum daily dose.
* age between 18 and 70
* voluntary and competent to consent

Exclusion Criteria:

* Major depressive disorder diagnosed with the DSM V criteria with a MADRS score >30 (actual)
* schizophrenia and other psychotic disorder
* drugs or alcohol abuse
* acutely suicidal
* significant head injury, or of any neurosurgical procedure with implanted material
* pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2015-03-12 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
score improvement on the Yale Brown Obsessive and Compulsive Scale after one month | 1 month after treatment
  % of improvement compare to baseline

SECONDARY OUTCOMES:
Number of responders on the YBOCS | 1 month after treatment
  Number of responders (decrease >35%) on the Yale Brown Obsessive and Compulsive Scale) or a score of 2 or less on the CGI-I (much or very much improved)
score improvement on the Yale Brown Obsessive and Compulsive Scale after 3 months | 3 months after treatment
  % of improvement compare to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bation Remy, MD, Principal Investigator — CH le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No